CLINICAL TRIAL: NCT07280663
Title: A Study on the Correlation Between the Level of Neurofilament Light Chain Protein and the Sensitivity to Remazolam in Older Adults
Brief Title: Correlation Between Neurofilament Light Chain and Remazolam Sensitivity in Elderly Adults
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: yuewei20251009
Record Dates: First submitted 2025-11-17; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Old Age
Keywords: old age; Neuronal filament light chain protein; Remazolane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with normal cognitive function (Experimental): MMSE scores tweney-seven or more points
  Interventions: Drug: Remazolane
- Group with declining cognitive function (Experimental): MMSE scores zero to twenty-seven
  Interventions: Drug: Remazolane

INTERVENTIONS:
Drug: Remazolane — Tramazolam via peripheral venous TCI is administered for sedation, with a concentration setting of 0.26 μg/mL. The infusion of tramazolam is stopped once the patient's consciousness has disappeared, which is indicated by the absence of eyelash reflex. The amount of tramazolam used, the time until consciousness disappeared, the time until awakening, and the BIS value are recorded.

SUMMARY:
With the acceleration of population aging, China has entered a stage of "deep aging." According to data from the Seventh National Census of Population released in 2021, the proportion of individuals aged 60 or older is 18.70%, with a total number of 264 million, while the proportion of individuals aged 65 or older is 13.50%, with a total number of approximately 190 million. As the proportion of elderly individuals continues to rise, the number of elderly patients undergoing surgical procedures has also increased significantly. Elderly individuals often suffer from multiple chronic diseases, a decline in physiological reserve function, and a reduced tolerance to anesthesia and surgery, presenting new challenges for anesthesiologists. Moreover, cognitive dysfunction is prevalent among the elderly and increases with age . Cognitive dysfunction before surgery is not only closely related to postoperative complications, delirium, further deterioration of cognitive function, and increased mortality, but also leads to longer hospital stays and higher medical expenses after surgery.Therefore, it is of great significance to timely and accurately identify whether the cognitive function of the elderly has been impaired and to actively implement targeted intervention strategies to maintain the health and prognosis of elderly surgical patients, as well as to control the social medical costs.

DETAILED DESCRIPTION:
1.1) To investigate the correlation between the levels of neurofilament light chain protein and the scores obtained from the Mini-Mental State Examination (MMSE).

2) Investigate the correlation between the levels of neurofilament light chain protein and the sensitivity to remazolam in elderly patients.

3) Study the factors that influence the sensitivity of remazolane in elderly patients.

2.Methods: One hundred and twenty-eight patients undergoing knee joint replacement were divided into normal cognitive group and cognitive decline group according to MMSE score.

3.MAIN OUTCOME MEASURES: (1) Age, gender, education level, BMI, ASA classification, smoking history, drinking history, cardiovascular disease history, diabetes mellitus history, hyperlipidemia history and COPD history. (2) BP, MAP, HR, degree of saturation of blood oxygen and BIS were measured after entering the room, after the level of spinal anesthesia was stable, when the patient lost consciousness (mascara reflex was lost) after the patient was injected with Rimazolam, and when the patient woke up immediately after the patient stopped taking the drug. (3) The time of consciousness loss (loss of eyelashes reflection) after the injection of rumazine, and the amount of drug injection. (4) How long the patient wakes after stopping the medication. (5) MMSE scores of patients. (6) Take 2 ml cerebrospinal fluid to measure NFL level.

4.The mean ± SD was used to express the measurement data. The difference between the two groups was analyzed by t-test. One-way analysis of variance (ANOVA) was used to compare the data between the two groups.The counting information is represented in examples (percentages) and the comparison of the rates between the two groups is based on a cartesian test. Multivariate Logistic regression analysis was used to analyze the determinants of sensitivity to RZL. The correlation between NFLP and sensitivity to RZL was analyzed by Superman correlation coefficient.P < 0.5 was significant difference.

ELIGIBILITY:
Inclusion Criteria:

* Elective knee joint replacements.
* Age ≥ 60 years.
* ASA rating I ~ III.

Exclusion Criteria:

* Persons who have recently used sedatives or opioids.
* Persons who are allergic to narcotic drugs.
* People with clotting disorder, infection at the site of the puncture, spinal deformities or spinal disorders.
* Those who have been diagnosed with nervous system disorders.
* Patients or family members refuse to participate in this study.
* Exit research for their own reasons.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
neurofilament light chain protein | 24 hours
  Differences in level of neurofilament light chain protein
Loss of consciousness time | 24hours
  Differences in loss of consciousness time
awakening time | 24 hours
  Differences in awakening time
Remazolane dosage | 24 hours
  Differences in Remazolane dosage
Mean Arterial Pressure (MAP) | 24 hours
  Differences in Mean Arterial Pressure (MAP)
heart rate | 24 hours
  Differences in heart rate
Electroencephalographic dual frequency index (BIS value) | 24 hours
  Differences in Electroencephalographic dual frequency index (BIS value)
Incidence of adverse effects (hypotension, bradycardia, respiratory depression) | 24 hours
  Incidence of adverse effects (hypotension, bradycardia, respiratory depression)

SECONDARY OUTCOMES:
Use of vasoactive drugs | 24 hours
  Use of vasoactive drugs

OTHER OUTCOMES:
Checklist form: Age, gender, education level, , ASA grade, smoking history, drinking history, cardiovascular disease , diabetes mellitus , hyperlipidemia, and COPD | 24 hours
BMI | 24 hours
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Second Hospital of Shanxi Medical University, Taiyuan, Shanxi, China